CLINICAL TRIAL: NCT01072032
Title: Cortical and Biomechanical Dynamics of Ankle Robotics Training in Stroke
Acronym: AbotMot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: A7251-W; HP-00043705 (Other: University of Maryland, Baltimore, IRB)
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Results first posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-05

CONDITIONS: Cerebral Stroke
Keywords: EEG; Robotics (ankle); Motor-learning; Brain Plasticity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-Reward (Experimental): Low-Reward Anklebot training Group: The low reward-feedback group receives the Anklebot training with only immediate feedback on target successes, without cumulative scores and with minimal social interaction with the research team.
  Interventions: Device: Anklebot (Ankle Robot)
- High-Reward (Active Comparator): High-Reward Anklebot training Group: The high-reward group receives cumulative scores and abundant social interaction and are eligible for prizes during each training session and at completion of the study
  Interventions: Device: Anklebot (Ankle Robot)

INTERVENTIONS:
Device: Anklebot (Ankle Robot) — Impedance controlled ankle robot provides assistance as needed for participants to perform ankle movements while playing a video game, is used to assist stroke patients to enhance motor recovery

SUMMARY:
Reduced mobility is often a long-term problem facing those who have chronic leg weakness resulting from stroke. Recent innovations in stroke therapy have applied motor learning principles to improve motor skills through regular practice of activities using the weaker limb. Because the ankle provides critical torques for normal walking and mobility function, impairments at the affected ankle pose a major limitation to achieving optimal mobility recovery. To address this we have developed a novel ankle robot (Anklebot) to enhance physical therapy for improving walking and mobility after stroke. This computer controlled device provides assistance when users cannot complete a movement, but will not assist if the user is active.

Motor learning requires active involvement in task-related practice to mediate brain plasticity. While voluntary movement is important to remodel motor control circuits, the brain mechanisms of reward and motivation also can play an important role. Core brain networks involved in reward and motivation increase a person's involvement with their surroundings, to focus attention and to prompt one to approach reward and avoid punishment. This increased involvement and the elevated emotions associated with it have been shown to enhance performance, memory and learning.

The purpose of this study is to investigate responses of brain and motor behavior of stroke patients who use the Anklebot during a 3-week / 3-session/week motor learning based training. These responses are compared to a 3-week delayed entry period in which the participants will perform an at-home walking program of equal time. After the 3-week delayed entry walking program, subjects are divided into low and high reward-feedback groups. The low reward-feedback group receives the Anklebot training with only immediate feedback on target successes, without cumulative scores and with minimal social interaction with the researchers. The high-reward group receives cumulative scores and ongoing social support, are eligible for prizes during each session and at the study's completion. All subjects play the games as noninvasive electroencephalography and electromyography record brain and muscle activity. In addition to analyzing brain information before and after the Anklebot training, ankle motor control and walking functions are also assessed immediately before and after the first and last robotic training sessions.

DETAILED DESCRIPTION:
After informed consent is obtained, this pilot study will require at least eleven visits for all subjects. The first visit will entail screening and eligibility tests that last about 3 hours and will occur at the VAMC (Veteran's Administration Medical Center) in the Geriatric Assessment Clinic (GAC). The second and third visits will last approximately 3 hours at the VAMC Human Motor Performance Laboratory and will involve collection of noninvasive EEG, surface EMG and ECG, and practice of ankle movements by using the ankle robot to play video games. In addition measures of gait and balance function will be assessed pre- and post- the Anklebot training. For the next 3-weeks the subjects will take part in an at-home, monitored (log) walking program. The next seven visits (the training program) entail further practice of ankle movements by using the ankle robot to play video games, collection of motor control data but not the collection of any electrophysiological data.. Visit eleven (final) is the same as visits 2 & 3.

Visit 1: Screening evaluations include review of medical records, medical and neurologic examinations to determine eligibility. Clinical evaluations will also include the Mini Mental State Exam (MMSE) and the Center for Epidemiologic Study (CES-D). Clinical suspicion or evidence on these screening instruments of dementia, depression, or other cognitive deficits that could interfere with the study will preclude further study evaluation and prompt referral to psychiatry or other appropriate health professional for further evaluation. The Automated Neuropsychological Assessment Metrics (ANAM) is also administered as a comprehensive neuropsychological tool for measuring multiple facets of neuropsychological processes that pertain to cognitive function and motor learning. In addition participants will be asked to walk 10 meters 3 times across a gait measuring mat at their preferred speed while in a safety harness and accompanied (not assisted) by an experienced research assistant. This will help determine their deficit severity for grouping during data analysis. Finally, a standard neurological examination is conducted by medically credentialed staff.

Visit 2 & 3 & 11: After study enrollment and medical screening, subjects will be tested with the Anklebot while EEG, EMG, and heart rate (ECG) are recorded.

First, subjects will be fitted with a stretch-lycra cap that houses 64 recessed EEG sensors formed from tin. The participant's skin will be lightly abraded or rubbed with the end of a Q-tip at each sensor site to remove oil and dead epidermal tissue to establish good conductance of the EEG signal. The skin will not be broken. Using a blunt applicator attached to a syringe, an FDA-approved non-toxic conducting gel will then be applied through an opening in each of the 64 recording sensors to establish continuous contact of the gel between the skin at the recording sites and the corresponding sensors. Recording sensors will also be positioned on the skin above and below the left eye to monitor eye movements as well as on both ear lobes to serve as "non-brain" reference sites. A ground electrode site will be applied in the frontal region. The eye-channel and reference sites will be lightly abraded with a pad, rubbed with alcohol, and prepared with the conducting gel to enable continuous connection between the scalp and the sensor surface. Also, surface EMG electrodes will be applied to tibialis anterior, gastrocnemius, and, if needed, the peroneal muscles of the paretic leg. Leads for ECG recording will be applied bilaterally to locations immediately inferior to the clavicles.

Once the set-up is complete, subjects will be asked to walk 10 m over an instrumented gait mat to record gait parameters during 3 preferred and 3 fastest walking trials. Subjects will be asked to repeat these walking tasks while performing a concurrent cognitive task consisting of solving and verbally reporting answers to simple arithmetic problems. They will wear a gait belt and be attended closely by research staff as they walk and receive seated rests as required to prevent fatigue. A second test will measure balance control by recording 30 second trials of postural sway during quiet standing on a force plate. Three balance conditions include eyes open, eyes closed, and eyes open while performing a concurrent cognitive task consisting of solving and verbally reporting answers to simple arithmetic problems. Seated rests will be provided as needed.

After baseline functional testing participants will be seated in a chair and the ankle robot will be attached to their paretic leg by means of an orthopedic knee brace and an orthopedic shoe. Pads and cushioning will be applied as needed for proper fitting, and the knee brace will be mounted to the chair for stability. The leg will rest on a cushioned support with the knee at 45 degrees and the foot free to move.

Once the set-up is completed, subjects will be asked to "play" a series of videogames by plantar- or dorsi-flexing the paretic ankle to move a corresponding cursor on a computer screen in order to hit slowly moving targets. The first game is about two-minutes duration and is played without robotic assistance to assess subjects' baseline motor control and ability. Subsequently, 6 games of about 4-minutes duration will provide differing levels of robotic support to guide or encourage the subjects to complete the prescribed ankle movements. The nature and amount of robotic support will be varied across the session to promote short-term motor learning and control of the paretic ankle. Upon completion of the performance-based training series, a repeat of the two-minute unassisted game completes the session.' Finally, subjects will be asked to repeat the postural sway and walking tests as before.

Visits 4-10: participants will be seated in a chair and the ankle robot will be attached to their paretic leg by means of an orthopedic knee brace and an orthopedic shoe. Pads and cushioning will be applied as needed for proper fitting, and the knee brace will be mounted to the chair for stability. The leg will rest on a cushioned support with the knee at 45 degrees and the foot free to move.

Once the set-up is completed, subjects will be asked to "play" a series of videogames by plantar- or dorsi-flexing the paretic ankle to move a corresponding cursor on a computer screen in order to hit slowly moving targets. The first game is about two-minutes duration and is played without robotic assistance to assess subjects' baseline motor control and ability. Subsequently, 6 games of about 4-minutes duration will provide differing levels of robotic support to guide or encourage the subjects to complete the prescribed ankle movements. The nature and amount of robotic support will be varied across the session to promote short-term motor learning and control of the paretic ankle. Upon completion of the performance-based training series, a repeat of the two-minute unassisted game completes the session. During these training sessions no electrophysiological data will be acquired, only motor control data acquired by the Anklebot itself.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke greater than 3 months prior
* Residual hemiparetic gait with observable asymmetry in the gait pattern.
* Women or men aged 21 to 85 years
* Completed all conventional physical therapy.
* Adequate language and neurocognitive function to participate in training, testing, and to give informed consent.
* Minimal ankle flexion in either direction (dorsi- or plantar-)

Exclusion Criteria:

* MMSE score < 23 (9th grade education or more) or MMSE score < 17 (8th grade education or less)
* CES-D score > 16
* Clinical history of orthopedic, chronic pain or severe neuromuscular disorders restricting participation in a short term ankle movement training paradigm.
* Severe or global receptive aphasia which confounds reliable testing and training.
* Women of child-bearing potential, if there is any self-reported chance that they may be pregnant.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-05; Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald N Goodman, PhD, Principal Investigator — VA Maryland Health Care System, Baltimore
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goodman RN, Rietschel JC, Roy A, Jung BC, Diaz J, Macko RF, Forrester LW. Increased reward in ankle robotics training enhances motor control and cortical efficiency in stroke. J Rehabil Res Dev. 2014;51(2):213-27. doi: 10.1682/JRRD.2013.02.0050. PMID 24933720

RESULTS

PARTICIPANT FLOW:
Groups:
- Low-Reward: Low-Reward Anklebot training Group
  Anklebot (Ankle Robot): Impedance controlled ankle robot provides assistance as needed for participants to perform ankle movements while playing a video game, is used to assist stroke patients to enhance motor recovery
- High-Reward: High-Reward Anklebot training Group
  Anklebot (Ankle Robot): Impedance controlled ankle robot provides assistance as needed for participants to perform ankle movements while playing a video game, is used to assist stroke patients to enhance motor recovery
Period: Overall Study
Arm/Group | Low-Reward | High-Reward
Started | 13 | 14
Completed | 5 | 5
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Reward | High-Reward | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 6 | 9 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (4.3) | 59.2 (5.4) | 60.5 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Motor Control
Description: Normalized jerk is a measure of movement smoothness, derived from jerk [(meters)/(second cubed)] divided by the peak velocity (meters/second), leaving values in units of 1/second squared (ie., 1/s^2)
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: 1/s^2
Groups:
- Low-Reward: Low-Reward Anklebot training Group
  Anklebot (Ankle Robot): The low reward-feedback group receives the Anklebot training with only immediate feedback on target successes, without cumulative scores and with minimal social interaction with the research team.
Arm/Group | Low-Reward | High-Reward
Number analyzed (Participants) | 5 | 5
1/s^2 | 413.22 (140.67) | 523.94 (152.02)

2. Secondary Outcome: Functional Walking Measures
Description: Preferred, self-selected walking velocity measured in centimeters/second (i.e., cm/s).
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Low-Reward | High-Reward
Number analyzed (Participants) | 5 | 5
cm/s | 89.45 (45.95) | 78.86 (40.06)

3. Secondary Outcome: EEG Spectral Coherence Estimates
Description: EEG coherence reflects the degree to which brain regions communicate. It is derived from calculating the degree of association between regions in specified frequency bandwidths; it is like a correlation, except that the values range from 0-1 instead of -1 to 1, so technically there are no units as it is a coefficient. Higher coherence values indicate stronger associations between regions.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: Coherence ratio
Arm/Group | Low-Reward | High-Reward
Number analyzed (Participants) | 5 | 5
Coherence ratio | .35 (.08) | .55 (.067)

ADVERSE EVENTS:
Time Frame: During the period of active enrollment in the study, covering initial intake screening, followed by 3 weeks of activity and post-testing: total 4-5 weeks.
Arm/Group | Low-Reward | High-Reward
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 2/13 | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Reward (N=13) | High-Reward (N=14)
Fall at home (Nervous system disorders) | 1 (1) | 1 (1) — Two participants fell during course of normal home life. These were deemed not to be study-related by Data Safety Monitoring Board
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Not study related. Participant placed on medical hold until cleared by physician.
Hip soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Participant complained of hip pain after early walking sessions. Withdrew from study due to other medical problems not study-related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes